CLINICAL TRIAL: NCT01274286
Title: Evaluation of the Effectiveness of the New Hospital Accreditation
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Che-Ming Yang, Department of Health Care Administration, Taipei Medical University
Other Study IDs: 99069
Record Dates: First submitted 2011-01-09; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Hospital Accreditation
Keywords: hospital accreditation; patient-centered; healthcare quality index; documentary analysis; meta analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Since the first hospital accreditation was implemented in our country in 1978, we have become the fifth in the world, the first in Asia that applied the system of hospital accreditation. While discussing the development of the hospital accreditation history of Taiwan, different concerns have been raised over time.

The main objective of this study is to scrutinize if there have been any quality improvement of healthcare that hospitals delivered since the renewal of hospital accreditation standards. Also, in order to provide suggestions to make the hospital accreditation a better one, this study firstly endeavors to locate the differences which were brought out by both the old and the new hospital accreditation.

Second, this study will analyze and survey the impacts of accreditation on hospitals' performance and healthcare. After finishing the first two steps, this study will then state updated improvement suggestions.

Documentary analysis and meta analysis will be the two major scientific research methods in this study. Data will be collected from various resources, such as government agencies, private research institution and hospitals around the nation. By collecting raw data broadly and deeply, the accountability, therefore, can be ensured.

Throughout the efforts of identifying differences between the new and old accreditation standards, comparing hospitals' scores on performance index and finding evidence of performance improvement, we hope this study would provide the most comprehensive and solid suggestions to improve our hospital accreditation system.

ELIGIBILITY:
Inclusion Criteria:

* above 20 years old

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients Doctors
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Che-Ming Yang, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan